CLINICAL TRIAL: NCT02955940
Title: An Open-Label, Multicenter, Rollover Study to Enable Continued Treatment Access for Subjects Previously Enrolled in Studies of Ruxolitinib
Brief Title: An Open-Label Study to Enable Continued Treatment Access for Subjects Previously Enrolled in Studies of Ruxolitinib
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-270; 2023-507225-42-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Colorectal Cancer (CRC); Breast Cancer; Lung Cancer
Keywords: Solid tumors; ruxolitinib; regorafenib; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Lung Neoplasms | interventions — ruxolitinib; Capecitabine; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ruxolitinib (Experimental): Study treatment for participants should be the same as the dosage from the parent study at the time the roll over protocol is initiated. Dose modifications are permitted.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib plus background cancer therapy (Experimental): Study treatment for participants should be the same as the dosage from the parent study at the time the roll over protocol is initiated. Dose modifications are permitted.
  Interventions: Drug: Ruxolitinib; Drug: Capecitabine; Drug: Regorafenib
- Background cancer therapy alone (Experimental): Capecitabine and Regorafenib at the same dose provided in the parent study at the time of the rollover.
  Interventions: Drug: Capecitabine; Drug: Regorafenib

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg BID
  Other Names: INCB018424; Jakafi®
  Arms: Ruxolitinib; Ruxolitinib plus background cancer therapy
Drug: Capecitabine — Capecitabine at the same dose provided in the parent study at the time of the rollover.
  Other Names: Xeloda®
  Arms: Background cancer therapy alone; Ruxolitinib plus background cancer therapy
Drug: Regorafenib — Regorafenib at the same dose provided in the parent study at the time of the rollover.
  Other Names: Stivarga®
  Arms: Background cancer therapy alone; Ruxolitinib plus background cancer therapy

SUMMARY:
The purpose of this study is to provide continued supply of ruxolitinib alone, ruxolitinib plus background cancer therapy, or background cancer therapy alone to subjects from an Incyte-sponsored study of ruxolitinib that has reached its study objectives or has been terminated.

This study will also provide another mechanism for reporting adverse events related to study drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled and receiving treatment in an Incyte-sponsored clinical study of ruxolitinib that has completed or been terminated.
* Currently tolerating treatment in the parent protocol.
* Currently benefiting from the treatment with ruxolitinib alone, ruxolitinib plus background cancer therapy, or background cancer therapy alone, as determined by the investigator.
* Have at least stable disease, as determined by the investigator.
* Has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements.

Exclusion Criteria:

* Has been permanently discontinued from study treatment in the parent study for any reason.
* Able to access ruxolitinib and/or background cancer therapy outside of the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and types of adverse events and serious adverse events | Maximum duration of every 2 months (maximum duration of 1 month for subjects receiving regorafenib) from enrollment through 30-37 days after end of treatment up to 24 months.
  Subjects will be treated until disease progression or discontinuation criteria are met.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (9):
- United States (6):
  - UCLA Healthcare Hematology-Oncology, Santa Monica, California
  - University of Louisville, Louisville, Kentucky
  - New York Oncology Hematology Pc., Clifton Park, New York
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical Consultants Llc, The Woodlands, Texas
- Poland (3):
  - Sp Zoz Szpital Uniwersytecki W Krakowie Oddzial Kliniczny Hematologii, Krakow
  - Samodzielny Publiczny Szpital Kliniczny, Lublin
  - Instytut Hematologii I Transfuzjologii, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: An Open-Label Study to Enable Continued Treatment Access for Subjects Previously Enrolled in Studies of Ruxolitinib — https://incyteclinicaltrials.com/studies/incb-18424-270